CLINICAL TRIAL: NCT06322329
Title: RealMove (Lung): Assessing Tumour Motion With Dynamic MRI
Acronym: RealMove(lung)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Collaborators: Uppsala University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K 2023-10103
Record Dates: First submitted 2024-03-08; First posted 2024-03-21 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-04

CONDITIONS: Lung Tumor
Keywords: Radiotherapy; Motion management; Dynamic MRI
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Full cohort (Experimental): All subjects are included in the same arm.
  Interventions: Other: Dynamic MRI

INTERVENTIONS:
Other: Dynamic MRI — Subjects receive a study-specific dynamic MRI scan. If the hypothesis of the study is confirmed, this examination can be used to inform future patients' treatment planning, replacing the use of 4D CT.

SUMMARY:
The study aims to develop an improved method to tailor the geometric safety margin when treating with stereotactic body radiotherapy (SBRT), to avoid tumour cells being missed during irradiation and to limit the exposure of normal tissues as much as possible. Dynamic magnetic resonance imaging (MRI) is assumed to represent the tumour motion during the respiratory cycle more realistically, compared to 4-dimensional computed tomography (4D CT), thanks to its high temporal resolution and the possibility to image the motion over a longer period of time. Patients receiving SBRT for a pulmonary target located below the level of the carina are included in the study, and the hypothesis will be tested through a comparison of the tumour amplitude measured with each modality. Furthermore, the predictive value of the image series acquired at treatment planning, for the motion patterns observed at each treatment fraction, will be evaluated through repeated 4D CBCT acquisitions.

DETAILED DESCRIPTION:
In the current study, a 2D-cine MRI examination will be performed, in addition to the 4D CT examination that is standard for patients receiving radiotherapy for tumours in the thorax or abdomen. A subgroup of the study participants (referred to as the 4D CBCT subcohort) will also be required to perform a 4D CBCT examination at three treatment sessions. The main cohort consists of 95 subjects and the 4D CBCT subcohort of 55 subjects. The study does not involve any change in the treatment routine; rather, the study images are collected for retrospective analysis. Following each imaging session, the subject should fill out an anxiety questionnaire and their pulse will be measured, to give an indication of any anxiety which might influence the breathing pattern of the current session.

Clinical follow-up will be performed retrospectively by reviewing the participants' medical records. Progress, health status and treatment-related toxicity will be evaluated, up to 10 years after completed treatment.

The study objectives are:

* To evaluate dynamic MRI for characterising the respiratory-related tumour motion, compared to the current standard modality of 4D CT.
* To evaluate the variation in breathing motion at different times points.
* To evaluate the clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Accepted for SBRT treatment of one or more caudally situated lung targets (NSCLC or metastases), i.e. below the carina.
* Age ≥ 18 years
* Adequate clinical condition to maintain immobilised position for at least 30 minutes
* Adequate Swedish skills and cognitive function to understand study information and to fill in the questionnaire

Exclusion Criteria:

* Pregnancy or breastfeeding, or planned pregnancy or breastfeeding, during treatment
* Contraindication for MRI examination
* Otherwise incapable of participating in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2026-03-17 (Estimated); Study Completion 2036-03-17 (Estimated)

PRIMARY OUTCOMES:
Difference in amplitude of the tumour motion, as assessed by dynamic MRI and 4D CT, respectively | Over 3-4 weeks: twice pre-treatment, and three times during treatment
  The two dynamic scans represent the tumour motion through different techniques. If the amplitude indicated by 4D CT is smaller than that indicated by dynamic MRI, the hypothesis is confirmed.
Difference in amplitude of the tumour motion, assessed at different times (using dynamic MRI and 4D CBCT) | Over 3-4 weeks: twice pre-treatment, and three times during treatment
  4D CBCT images are acquired at each treatment session, in treatment position. These will assess the stability of the breathing patter through the treatment course.
Difference in the structure of the probability density function, assessed at different times | Over 3-4 weeks: twice pre-treatment, and three times during treatment
  The breathing pattern is represented by a probability density function, indicating the regularity of the motion. The stability of this pattern through the treatment course will be assessed.

SECONDARY OUTCOMES:
Anxiety during examinations of tumour motion | Over 3-4 weeks: twice pre-treatment, and three times during treatment
  Measured by a questionnaire
Overall survival | Up to 10 years after treatment
  Review of medical records
Progression-free survival | Up to 10 years after treatment
  Review of medical records
Grade ≥2 toxicity assessed by CTCAE v.5.0 | Up to 10 years after treatment
  Review of medical records

CONTACTS AND LOCATIONS:
Overall Officials: Eva Onjukka, PhD, Principal Investigator — Karolinska University Hospital/Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden